CLINICAL TRIAL: NCT00684268
Title: Multicenter Study To Evaluate The Efficacy Of Silymarin In Addition To Combination-Therapy With Pegylated Interferon Alfa 2a (Peg-Ifn Alfa 2a) And Ribavirin In Patients With Chronic Hepatitis C
Brief Title: Intravenous Silibinin in Combination With Peg-interferon and Ribavirin in Nonresponders
Acronym: NRSily
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Peter Ferenci, Prof. of Medicine, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRSili
Record Dates: First submitted 2008-05-19; First posted 2008-05-26 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C
Keywords: silibinin; chronic hepatitis C; peginterferon; ribavirin; nonresponders; efficacy of iv. silibinin; safety
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — Silybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- on treatment nonresponders (Experimental): naive patients with null response to peginterferon/ribavirin at week 12 or partial response at week 24
  Interventions: Drug: Silibinin
- Nonresponders to previous antiviral combination therapy (Experimental): Nonresponders defined by viral status at weeks 4,12, and 24 of previous peginterferon/ribavirin combination therapy
  Interventions: Drug: Silibinin

INTERVENTIONS:
Drug: Silibinin — comparison of different dosing schedule of Silibinin infusions (20 mg/kg/d infused over 2 hours) A: 3x5days B: 14 days C: 21 days D: 28 days
  sequential the infusion duration will be shortened - 2 hours, then 1 hr and then 1/2 hr/infusion
  Other Names: Silibinin infusions (20 mg/kg/d infused over 2 hours)given for 21 (either Monday -Friday or daily) or 28 days, continuation of antiviral combination therapy
  Arms: Nonresponders to previous antiviral combination therapy
Drug: Silibinin — 20 mg/kg Silibinin iv /d /21 days, antiviral combination therapy will be continued
  Arms: on treatment nonresponders

SUMMARY:
By chance the investigators found that iv. silibinin has a potent antiviral effect against the hepatitis C virus. Based on the results of the dose finding study (published) te optima dosing schedule is explored.This study will be evaluate whether the highest active dose given for the optimal time combined with standard of care will result in a sustained virologic response (=cure of hepatitis C).

DETAILED DESCRIPTION:
Since the publication of the first data the optimal dosing schedule is investigated

ELIGIBILITY:
Inclusion Criteria:

* Nonresponders to full dose PEG-IFN/RBV therapy
* Liver biopsy within the last 2 year

Exclusion Criteria:

* Intolerance to one of the study drugs
* Coinfection with HIV/HBV

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-10; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
viral response at week 24 | week 24

SECONDARY OUTCOMES:
sustained virologic response | week 72
Safety | week 72
  start to end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Beinhardt S, Rasoul-Rockenschaub S, Scherzer TM, Ferenci P. Silibinin monotherapy prevents graft infection after orthotopic liver transplantation in a patient with chronic hepatitis C. J Hepatol. 2011 Mar;54(3):591-2; author reply 592-3. doi: 10.1016/j.jhep.2010.09.009. Epub 2010 Oct 14. No abstract available. PMID 21106270
- [Result] Ferenci P, Scherzer TM, Kerschner H, Rutter K, Beinhardt S, Hofer H, Schoniger-Hekele M, Holzmann H, Steindl-Munda P. Silibinin is a potent antiviral agent in patients with chronic hepatitis C not responding to pegylated interferon/ribavirin therapy. Gastroenterology. 2008 Nov;135(5):1561-7. doi: 10.1053/j.gastro.2008.07.072. Epub 2008 Aug 3. PMID 18771667
- [Result] Payer BA, Reiberger T, Rutter K, Beinhardt S, Staettermayer AF, Peck-Radosavljevic M, Ferenci P. Successful HCV eradication and inhibition of HIV replication by intravenous silibinin in an HIV-HCV coinfected patient. J Clin Virol. 2010 Oct;49(2):131-3. doi: 10.1016/j.jcv.2010.07.006. Epub 2010 Aug 14. PMID 20709593
- [Result] Rutter K, Scherzer TM, Beinhardt S, Kerschner H, Stattermayer AF, Hofer H, Popow-Kraupp T, Steindl-Munda P, Ferenci P. Intravenous silibinin as 'rescue treatment' for on-treatment non-responders to pegylated interferon/ribavirin combination therapy. Antivir Ther. 2011;16(8):1327-33. doi: 10.3851/IMP1942. PMID 22155914